CLINICAL TRIAL: NCT03407690
Title: A Study to Assess the Carriage of Pneumococci in Children Aged ≤8 Years, and Their Household Contacts
Acronym: PIN2
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: PIN2
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2018-08

CONDITIONS: Immunization; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PIN2 study participants: All those giving swabs for the study
  Interventions: Other: nasal swab

INTERVENTIONS:
Other: nasal swab — collection of nasal swab to allow carriage of pneumococci to be assessed

SUMMARY:
Since the introduction of pneumococcal conjugate vaccines, this research group has conducted several carriage studies. These were at key points in the evolution of the pneumococcal immunisation schedule, with regard to the introduction of PCV7, the change to PCV13 and the impending change in number of doses of PCV13 given to infants. The last carriage study, conducted in 2015/16 identified interesting changes in carriage patterns which will further be explored by the current planned study.

Nasopharyngeal swabs and saliva swabs will be taken from healthy subjects and any pneumococci present will be cultured and serotyped using standard methods, as per our previous studies (Hussain et al., 2005; Flasche et al., 2011; van Hoek et al., 2014).

DETAILED DESCRIPTION:
Streptococcus pneumoniae frequently colonises the human nasopharynx and most carriers remain asymptomatic. However, sometimes the organism may spread locally to cause non-invasive, mucosal infections such as sinusitis and otitis media or may invade the bloodstream and cause serious infections, including septicaemia, meningitis and pneumonia. In the 2005/06 epidemiological year, there were 6,391 cases of invasive pneumococcal diseases in England and Wales, with the highest incidence in the first year of life. The risk of developing invasive disease is dependent on both the susceptibility of the host and the invasiveness of the pneumococcus, which is largely determined by the characteristics of its polysaccharide capsule. Of the >90 known pneumococcal serotypes, the seven serotypes (4, 6B, 9V, 14, 18C, 19F and 23F) included in the 7-valent pneumococcal conjugate vaccine (PCV7) accounted for around 75% of childhood IPD cases in England and Wales prior to routine pneumococcal vaccination.

There have been several carriage studies conducted by this group at key points in the evolution of the pneumococcal vaccination policy of the UK, before use of any PCV, once the PCV7 had been introduced and once the change to PCV13 had been made. Studies have shown that conjugate vaccines, of which PCV7 and PCV13 are examples, can affect carriage of the bacteria against which the vaccinate. This series of carriage studies is important in understanding which pneumococcal strains are in the nose and so are potentially part of the chain of transmission as the vaccinations given have changed. For pneumococcus, where there are many strains, it is important to understand whether clearing carriage of a strain contained in the vaccine creates a niche which can be exploited by a strain of greater virulence or one which causes more serious disease. Our last such study suggested there are changes which we should continue to monitor, which is why the current study is now happening.

Nasopharyngeal swabs and saliva swabs will be taken from healthy subjects and any pneumococci present will be cultured and serotyped using standard methods, as per our previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. At least one child aged ≤8 years in the household
2. Written informed consent obtained from the child's parent / legal guardian for their participation, and for any participating household contacts

Exclusion Criteria:

* Moderate to severe cerebral palsy or other debilitating condition
* Syndromes and neurological disorders affecting swallowing.
* Ear, nose & throat disorders affecting local anatomy for swabbing (e.g. malformed ears)
* Confirmed or suspected immunodeficiency (congenital or acquired) or receiving immunosuppressive therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: • At least 200 children (index cases) aged ≤8 years and at least 200 household contacts.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
pneumococcal carriage rates | through study completion, expected 6 months
  pneumococcal carriage rates for PCV13 and non-PCV13 serotypes in children and infants eligible for primary or booster immunisation with PCV 13 and their household contacts

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD, Study Director — Public Health England
Locations (2):
- United Kingdom (2):
  - Gloucestershire Primary Care, Gloucester, Gloucestershire
  - Hertfordshire primary care, Hertford, Hertfordshire

IPD SHARING:
Plan to Share IPD: No